CLINICAL TRIAL: NCT03975192
Title: Efficacy of Neurostimulation on Opiate Withdrawal Symptoms in Pediatric ICU Patients
Brief Title: Neurostimulation for Opiate Withdrawal in the PICU
Acronym: NOW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no enrollment.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Karen Marcdante, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1185104
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Opiate Withdrawal Syndrome
Keywords: Opiate Withdrawal; Neurostimulation; Percutaneous Electric Nerve Field Stimulation; Pediatrics; Pediatric Intensive Care Unit

STUDY DESIGN:
Intervention Model Description: Study subject will be randomized to receive study treatment (PENFS device treatment) or the Standard of Care treatment (Methadone wean) for prevention of opiate withdrawal symptoms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): 50% of subjects will be randomized to the Intervention group and will receive percutaneous electric nerve field stimulation (PENFS) through the BRIDGE Device for 120 hours to treat withdrawal symptoms in patients following opiate exposure in the PICU.
  Interventions: Device: Percutaneous Electrical Nerve Field Stimulation
- Standard of Care Group (No Intervention): 50% of subjects will be randomized to the Standard of Care group and will receive be started on the standardized PICU Methadone wean for patients following opiate exposure in the PICU.

INTERVENTIONS:
Device: Percutaneous Electrical Nerve Field Stimulation — Placement of the PENFS device immediately following the last scheduled opiate dose in the PICU with active stimulation for 120 hours.
  Other Names: BRIDGE Device
  Arms: Intervention Group

SUMMARY:
This is a prospective pilot study to investigate the effects of Percutaneous Electrical Nerve Field Stimulation (PENFS) on symptoms of opioid withdrawal in pediatric patients in the intensive care unit.

DETAILED DESCRIPTION:
This is a prospective, unblinded, randomized controlled pilot trial to evaluate the impact of the BRIDGE device when used on patients at high risk of opioid withdrawal following opioid exposure.

The investigator team hypothesized that treatment of pediatric intensive care unit (PICU) patients (ages 5-17 years) with PENFS will prevent the development of opioid withdrawal symptoms, reduce the need for long-acting opioid agonists or pharmacological rescue agents to treat withdrawal, and decrease overall PICU length of stay (LOS).

Aim 1: Withdrawal, using the Withdrawal Assessment Tool (WAT-I) is less for those using PENFS device than for those receiving standard of care (SOC) treatment.

H1: The WAT-I will be lower in the PENFS group than the SOC group and this will be true, even after adjusting for age and total opioid dose/kg pre-weaning.

Aim 2: For withdrawal symptoms of nausea, vomiting or pain, those receiving PENFS compared to SOC will require less treatment for these symptoms.

H2: The PENFS groups compared to the SOC will have primarily fewer episodes of gastrointestinal distress and lower pain scores resulting in the use of fewer doses of rescue medications; further this will be true after adjusting for total opioid dose/kg pre- weaning.

Aim 3: PICU LOS will be less for those receiving the PENFS device compared to those receiving SOC treatment.

H3: Following the initiation of weaning, the PICU LOS will be less for those with PENFS than those with SOC. This will be true after adjusting for age and total opioid dose/kg pre-weaning.

The following inclusion and exclusion criteria will be used to determine eligibility for this study:

Inclusion:

* Children aged 5 to 17 years
* Admission to PICU at Children's Hospital of Wisconsin (CHW)
* Exposure to at least 120 hours of continuous IV opioid administration.

Exclusion:

* Age children <5 years
* Known central nervous system injury (hypoxic ischemic injury, traumatic brain injury, postoperative craniotomies),
* Plan to wean benzodiazepine dosing during the active study period
* Patients who are developmentally delayed
* Defined as inappropriately non-verbal for age and determined through review of the medical record and discussion with the PICU attending and consulting team members.
* Known pregnancy
* Any pregnancy testing done during the subject's hospitalization will be reviewed.

(This will only be monitored if required as SOC, but will not be collected for the purpose of the study alone.)

* Known seizure disorder
* Known diagnosis of psoriasis or significant dermatological disease involving ear (?)
* Patients with implantable devices (cardiac pacemaker, vagal nerve stimulator, etc.)

After consent, and prior to the initiation of opiate withdrawal initiation, subjects will be randomized to receive the local standard methadone wean or placement of the BRIDGE device. Randomization will be used to balance age (5-9 yrs., >9 yrs.) and gender (male, female) assigning subjects in a 1:1 ratio to the Bridge device or control groups.

Subjects in the treatment group will have the device placed immediately following their last scheduled opiate dose. The device will be active continuously for 120 hours from the time of placement. As needed (PRN) dosing of pain medication will be available for breakthrough symptoms experienced by the subject. Subjects randomized to the SOC group will begin SOC treatment per the PICU withdrawal protocol.

The BRIDGE device will be placed per manufacturer protocol. Electrodes will be placed percutaneously in the external ear with the help of a transilluminator to visualize the neurovascular bundles; three electrodes will be placed on the ventral and one on the dorsal aspect of the ear. The electrodes will be taped and secured behind the ear next to the generator itself which is secured to the skin with adhesive.

The electrode/needle arrays are placed according to the individual's distribution of neurovascular bundles. The exact location of the placement will vary slightly from person to person and is determined by both knowledge of auricular neuro-anatomy and visualization of the neurovascular bundles by transillumination (IHS, Versailles, IN, USA). The points will be targeted by four-point electrical stimulation using the BRIDGE device after carefully disinfecting the ear. The contents of the Neurostimulation will be delivered below sensation threshold for 5 consecutive days (120 hours).

Removal of the device will be done by a member of the study team if the patient is still admitted to CHW, or by the subject's parents if discharge takes place prior to the completion of the PENFS treatment. The device will be placed in a sharps discard container after removal. Subjects who will be discharged with the device will be provided with a sharps disposal bag that can be used to hold the device after removal. This bag can be discarded in any sharps container accessible to the subject or brought back to CHW and discarded the time of their next follow up appointment. If the subject's family is not comfortable removing the device at home the study team will make arrangements for the family to return to CHW for device removal.

If a patient in the PENFS group is experiencing significant breakthrough withdrawal symptoms (consistent WAT-I score of >4) for more than 48 hours, the PI and care team will meet to discuss whether scores are due to withdrawal symptoms or are being artificially inflated due to confounding factors. If the patient is determined to be experiencing significant symptoms of withdrawal, the device will be removed early, and the subject will be transitioned to SOC withdrawal treatment. At that point the patient will be considered to have withdrawn from study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 17 years
* Admission to PICU at Children's Hospital of Wisconsin (CHW)
* Exposure to at least 120 hours of continuous IV opioid administration.

Exclusion Criteria:

* Age children <5 years
* Known central nervous system injury (hypoxic ischemic injury, traumatic brain injury, postoperative craniotomies),
* Plan to wean benzodiazepine dosing during the active study period
* Patients who are developmentally delayed

  o Defined as inappropriately non-verbal for age and determined through review of the medical record and discussion with the PICU attending and consulting team members.
* Known pregnancy

  o Any pregnancy testing done during the subject's hospitalization will be reviewed. This will only be monitored if required as SOC, but will not be collected for the purpose of the study alone.
* Known seizure disorder
* Known diagnosis of psoriasis or significant dermatological disease involving ear (?)
* Patients with implantable devices (cardiac pacemaker, vagal nerve stimulator, etc.)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Withdrawal Assessment Tool (WAT-1) Score | Study Day 0 through Study Day 5
  Measurement of opiate withdrawal symptoms experienced by study subjects

SECONDARY OUTCOMES:
Pain Medication Use | Study Day 0 through Study Day 5
  Total dose of pain medications used on each study day
Pain Scores | Study Day 0 through Study Day 5
  Age appropriate pain score values for each study day
Length of Stay | PICU Admission
  Time PICU Admission to medical PICU discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No